CLINICAL TRIAL: NCT04983875
Title: Enhancing the Public Health Benefits of Mammography Screening by Informing Women of Both Breast Cancer and Breast Arterial Calcification Results: A Randomized Trial to Promote Cardiovascular Health
Brief Title: Mammography and Breast Arterial Calcification: An Information-Sharing Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Guy Montgomery, Professor, Department of Population Health Science and Policy, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: Study-21-00112; R01CA251754 (NIH)
Record Dates: First submitted 2021-07-22; First posted 2021-07-30 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-09

CONDITIONS: Mammography; Vascular Calcification
Keywords: Mammography; Breast Arterial Calcification; Women's Health; Preventive Medicine; Behavioral Medicine; Screening
MeSH Terms: conditions — Vascular Calcification

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BAC-enhanced group (Experimental): 944 participants will receive a post-mammography results letter which includes information on their BAC results.
  Interventions: Behavioral: BAC-Enhanced Letter
- Waitlist control group (Other): 944 participants will receive a post-mammography results letter without BAC information, which is the current standard of care. These patients will receive BAC information following study completion (approximately 6 months after mammography).
  Interventions: Behavioral: BAC-Enhanced Letter; Behavioral: Waitlist Control

INTERVENTIONS:
Behavioral: BAC-Enhanced Letter — The BAC-Enhanced Letter intervention includes enhancing the standard mammography results letter with a few additional lines of text informing patients of their personal BAC status.
Behavioral: Waitlist Control — Patients randomized to this group will receive a standard post-mammography results letter which does not include any information about their personal BAC status. However, participants randomized to this group will be informed of their personal BAC findings at the end of their study participation (approximately 6 months after mammography).
  Arms: Waitlist control group

SUMMARY:
The purpose of this research study is to determine the potential benefits of adding information on patients' breast arterial calcification (BAC) results to the standard results letter women receive after mammography. In addition to looking for potential breast cancer, research shows that mammograms can also detect the presence of calcifications within the breast arteries. Those calcifications can be associated with coronary artery disease. Right now, women are not routinely told whether or not they have BAC; that is, it's not part of standard practice to communicate that information to patients. However, previous research has suggested that patients would like to be informed about their BAC status more often. In this study, the team has two goals. First, the team wants to measure the rates of BAC in a large, representative group of 3,700 women.

Second, the study team wants to understand the effects of giving women information on their BAC results as part of their standard post-mammography letter. Specifically, the study team wants to see how sharing that information might affect women's healthcare choices and lifestyle. The research will include 400 women in this second part of the study, which will be the first in the literature to explore women's reactions to BAC information. If research shows that women find the information useful, BAC information may be given to women regularly in the future.

ELIGIBILITY:
Inclusion Criteria

* Female
* Scheduled to undergo mammography at one of Mount Sinai's breast radiology clinics (e.g., Dubin Breast Center, Radiology Associates)
* Age ≥ 40 years
* Read and speak English or Spanish
* Ability to understand and the willingness to sign a written informed consent
* Willing to sign and date any applicable medical record release documents for the study

Exclusion Criteria:

* Participants with known coronary artery disease (via self-report)
* Previous physician-diagnosed heart attack, stroke or TIA, heart failure, angina or taking nitroglycerin, or atrial fibrillation (via self-report or review of EMR)
* Inability to understand and comply with the instructions of the study due to the presence of cognitive or psychiatric conditions (such as dementia, psychosis, or mania), compromising ability to provide informed consent and/or follow study procedures
* Pregnant women

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 37000 (Estimated)
Dates: Start 2021-09-29 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Attendance at a cardiovascular appointment | Month 6
  Patients will be asked a YES/NO question asking them to report whether they have seen a healthcare provider to talk about their heart or coronary artery disease in the last six months. Patient's self-report responses will be confirmed via medical record review.

SECONDARY OUTCOMES:
Healthy Heart Score | Baseline
  The Healthy Heart Score is a survey to assess patients' heart healthy behaviors. It assesses age, smoking, body mass index, exercise, alcohol, and a composite diet score. A higher score indicates a greater risk of cardiovascular disease.
  Score has gender-specific algorithm that estimates 20-year CVD risk (https://healthyheartscore.sph.harvard.edu/) (DOI: 10.1161/JAHA.114.000954):
  20-yr CVD risk (%) "Healthy Heart Score" = [1 - 0. 9660 (exp [W- 6.57301)] × 100% where W= 0.10820 x age + 0.15285 (if past smoker) + 0.90138 (if current smoker) + 0.04676 × BMI - 0.01923 × g/d of alcohol + 0.0004 × (g/d of alcohol)2- 0.029251 × hrs/wk of physical activity - 0.05113 × diet score* 20-yr CVD risk (%) "Healthy Heart Score" = [1 - 0. 96368 (exp [W-7.2437)] × 100% where W= 0.13580 x age- 0.0005 x (age)2 + 0.06979 (if past smoker) + 0.42305 (if current smoker) +0.07424 × BMI - 0.00898 × g/d of alcohol + 0.0001 × (g/d of alcohol)2- 0.01755 × hrs/wk of physical activity - 0.06691 × diet score
Healthy Heart Score | Week 1
  The Healthy Heart Score is a survey to assess patients' heart healthy behaviors. It assesses age, smoking, body mass index, exercise, alcohol, and a composite diet score. A higher score indicates a greater risk of cardiovascular disease.
  Score has gender-specific algorithm that estimates 20-year CVD risk (https://healthyheartscore.sph.harvard.edu/) (DOI: 10.1161/JAHA.114.000954):
  20-yr CVD risk (%) "Healthy Heart Score" = [1 - 0. 9660 (exp [W- 6.57301)] × 100% where W= 0.10820 x age + 0.15285 (if past smoker) + 0.90138 (if current smoker) + 0.04676 × BMI - 0.01923 × g/d of alcohol + 0.0004 × (g/d of alcohol)2- 0.029251 × hrs/wk of physical activity - 0.05113 × diet score* 20-yr CVD risk (%) "Healthy Heart Score" = [1 - 0. 96368 (exp [W-7.2437)] × 100% where W= 0.13580 x age- 0.0005 x (age)2 + 0.06979 (if past smoker) + 0.42305 (if current smoker) +0.07424 × BMI - 0.00898 × g/d of alcohol + 0.0001 × (g/d of alcohol)2- 0.01755 × hrs/wk of physical activity - 0.06691 × diet score
Healthy Heart Score | Month 6
  The Healthy Heart Score is a survey to assess patients' heart healthy behaviors. It assesses age, smoking, body mass index, exercise, alcohol, and a composite diet score. A higher score indicates a greater risk of cardiovascular disease.
  Score has gender-specific algorithm that estimates 20-year CVD risk (https://healthyheartscore.sph.harvard.edu/) (DOI: 10.1161/JAHA.114.000954):
  20-yr CVD risk (%) "Healthy Heart Score" = [1 - 0. 9660 (exp [W- 6.57301)] × 100% where W= 0.10820 x age + 0.15285 (if past smoker) + 0.90138 (if current smoker) + 0.04676 × BMI - 0.01923 × g/d of alcohol + 0.0004 × (g/d of alcohol)2- 0.029251 × hrs/wk of physical activity - 0.05113 × diet score* 20-yr CVD risk (%) "Healthy Heart Score" = [1 - 0. 96368 (exp [W-7.2437)] × 100% where W= 0.13580 x age- 0.0005 x (age)2 + 0.06979 (if past smoker) + 0.42305 (if current smoker) +0.07424 × BMI - 0.00898 × g/d of alcohol + 0.0001 × (g/d of alcohol)2- 0.01755 × hrs/wk of physical activity - 0.06691 × diet score
Detection of coronary artery disease (CAD) | Month 6
  Participants will respond to a single, self-report item (adapted from the 2019 NHIS survey item) which will ask if they have been told by a doctor or other health professional that they had coronary artery disease in the last 6 months. The item will be rated as, "yes, no, or don't know." Self-reported diagnosis will be confirmed via medical record review.
Revised Illness Perception Questionnaire (IPQ-R) | Week 1
  Illness representations will be assessed using the IPQ-R which have been adapted to include an addendum of Cardiovascular-Disease Related Worry Scale questions. Participants will be asked to rate items related to personal beliefs about CAD with regard to causal beliefs and on 8 subscales: identity (scale 0-13); timeline (scale 6-30); consequences (scale 6-30); personal control (scale 6-30); treatment control (scale 5-25); illness coherence (scale5-25); timeline cyclical (scale 4-20); and emotional representations (scale 6-30); and CVD related worry scale (scale3-13). Full scale from 41-216, higher scores represent a higher number of symptoms related to CAD, more positive beliefs about the controllability of disease, and a greater personal understanding of the condition.
Revised Illness Perception Questionnaire (IPQ-R) | Month 6
  Illness representations will be assessed using the IPQ-R which have been adapted to include an addendum of Cardiovascular-Disease Related Worry Scale questions. Participants will be asked to rate items related to personal beliefs about CAD with regard to causal beliefs and on 8 subscales: identity (scale 0-13); timeline (scale 6-30); consequences (scale 6-30); personal control (scale 6-30); treatment control (scale 5-25); illness coherence (scale5-25); timeline cyclical (scale 4-20); and emotional representations (scale 6-30); and CVD related worry scale (scale3-13). Full scale from 41-216, higher scores represent a higher number of symptoms related to CAD, more positive beliefs about the controllability of disease, and a greater personal understanding of the condition.

CONTACTS AND LOCATIONS:
Overall Officials: Guy H. Montgomery, Ph.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There currently isn't a plan to share individual participant data (IPD) with other researchers as this is a single-center trial and all study investigators and personnel are affiliated with Mount Sinai.